CLINICAL TRIAL: NCT02937389
Title: Endoscopic Evaluation for Predicting the Complications Related to Gastric Conduit After Esophagectomy
Status: Completed | Type: Observational
Sponsor: Nagasaki University (Other)
Responsible Party: Principal Investigator, Kobayashi Shinichiro, Principal Investigator in department of Surgery, Nagasaki University
Other Study IDs: 16082202
Record Dates: First submitted 2016-10-17; First posted 2016-10-18 (Estimated); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Esophageal Neoplasms; Constriction; Anastomotic Leak; Ischemia
MeSH Terms: conditions — Esophageal Neoplasms; Constriction, Pathologic; Anastomotic Leak; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — dmpDNA
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Diagnostic Test: Patients after esophagectomy — Endoscopic examinations are performed at 1 and 8 postoperative days. Endoscopic examination is added when abnormal findings are demonstrated.

SUMMARY:
Gastric conduit ischemia or anastomotic breakdown after esophagectomy with cervical esophagogastrostomy often cause severe complications, such as leakage, necrotic organs, and strictures. Thus, the purpose of this study is the safety and efficacy of endoscopic evaluation about reconstructive organs after esophagectomy. The investigators evaluate endoscopic predictions using classifications in acute phase after esophagogastrostomy.

DETAILED DESCRIPTION:
The development and improvement of thoracoscopic esophagectomy (TE) reduced the severe pulmonary complication after esophagectomy. However, the postoperative complications relative to gastric conduit reconstruction are still common issues after esophagectomy. The ischemia of the proximal portion of the graft predisposes these patients to a high incidence of anastomotic complications after esophagectomy. Less commonly, severe graft ischemia can lead to transmural necrosis. Thus, early diagnosis of ischemic reaction may provide the suitable postoperative management and therapeutic intervention to prevent leakage, strictures and necrosis. Thus, the purpose of this study is the safety and efficacy of endoscopic evaluation about reconstructive organs after esophagectomy. The investigators evaluate endoscopic predictions using classifications in acute phase after esophagogastrostomy.

ELIGIBILITY:
Inclusion Criteria:

- Malignant or end-stage benign esophageal disease. Esophagectomy with reconstruction by a gastric pull-up.

Exclusion Criteria:

- Severe heart failure and pulmonary dysfunction Severe renal and liver dysfunction Allergenic history Pregnancy

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergo an esophagectomy with reconstruction by a gastric pull-up for malignant or end-stage benign esophageal disease. The patients have a cervical esophagogastrostomy.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-05; Primary Completion 2018-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
The classification of gastric conduit ischemia by endoscopic findings predicts the major complications of gastric conduit (strictures, leakage, necrosis) | From 1 to 29 days after esophagectomy

SECONDARY OUTCOMES:
Biological examination of the mucosal biopsy of gastric conduit as assessed by the ischemia related RNA copy number | From 1 to 15 days after esophagectomy
Biological examination of the mucosal biopsy of gastric conduit as assessed by the scoring system for immunohistochemical staining | From 1 to 15 days after esophagectomy
  The scoring system refer to the article entitled a scoring system for immunohistochemical staining: consensus report of the task force for basic research of the European Organization for Research and Treatment of Cancer-Gynaecological Cancer Cooperative Group
Biological examination of gastric conduit as assessed by the Mitochondrial DNA copy number | From 1 to 15 days after esophagectomy

CONTACTS AND LOCATIONS:
Overall Officials: Shinichhiro Kobayashi, M.D., Study Director — Nagasaki University Graduate School of Biomedical Sciences
Locations (1):
- Nagasaki University Hospital, Nagasaki, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kobayashi S, Kanetaka K, Yoneda A, Yamaguchi N, Kobayashi K, Nagata Y, Maruya Y, Yamaguchi S, Hidaka M, Eguchi S. Endoscopic mucosal ischemic index for predicting anastomotic complications after esophagectomy: a prospective cohort study. Langenbecks Arch Surg. 2023 Jan 17;408(1):37. doi: 10.1007/s00423-023-02783-x. PMID 36648542